CLINICAL TRIAL: NCT04158752
Title: Anti-CGRP Neutralizing Antibody for Modulation of Neurogenic Inflammation in Trigeminal and Glossopharyngeal Pain Associated With Small Fiber Neuropathy/Fibromyalgia
Brief Title: Anti-CGRP for Inflammation and Pain Modulation in Small Fiber Neuropathy/Fibromyalgia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103776
Record Dates: First submitted 2019-10-30; First posted 2019-11-12 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Trigeminal Neuralgia; Glossopharyngeal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia; Glossopharyngeal Nerve Diseases | interventions — galcanezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label Galcanezumab (Experimental): Participants will receive their 1st injectable dose during the Day 30 visit. Participants will then inject themselves at home on Day 60 and again on Day 90.
  Interventions: Drug: Galcanezumab

INTERVENTIONS:
Drug: Galcanezumab — Injection of study drug at 3 timepoints (day 30, day 60, day 90)

SUMMARY:
The investigators will treat patients (targeting enrollment of n=20) who suffer from trigeminal or glossopharyngeal nerve pain in the context of painful small fiber neuropathy. The primary pain-related objective is reduction of pain and reduced use of rescue and other anti-pain medications. Another goal is to monitor and confirm the safety profile established in the migraine population, during previous Phase 3 trials.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old.
* The patient must have an assigned diagnosis of non-neuralgic trigeminal nerve pain G50.1, with all its permutations listed in the ICD10 explicitly allowed. Co-morbid trigeminal neuralgia G50.0 and G43. … related headache codes are allowed. As an alternative to trigeminal nerve pain G50.1, glossopharyngeal nerve pain will be another inclusion criterion, with a G52.1 diagnosis and explicit mentioning of pain mediated by or in the innervation territory of the glossopharyngeal nerve.

In addition, patients have to be diagnosed with a painful small fiber neuropathy. This diagnosis is based on a skin biopsy or biopsy of an innervated surface epithelium with nerve fiber density count. The required ICD10 diagnostic codes are G63.3, G60.8, G62.8. Co-morbidity with a fibromyalgia-related disorder will be allowed, typically summarized under a diagnosis code of M79.7.

Exclusion Criteria:

* Patients that have a history of allergy or allergy-like incompatibility with a biologic that contains a human or humanized monoclonal antibody will be excluded.
* Female patients of child-bearing age who are or want to become pregnant will be excluded. In case such a patient intends to participate, then she has to commit to a pregnancy prevention regimen that is based on hormonal contraceptive or intra-uterine device.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sweta Sengupta, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral from a tertiary medical center. The first participant was enrolled July 24, 2020, and last participant was enrolled June 28, 2022.
Pre-assignment Details: Of the 26 enrolled, 20 patients met inclusion criteria.
Period: Overall Study
Arm/Group | Open Label Galcanezumab
Started | 20
Completed | 18
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Galcanezumab
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (12.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Score
Description: Patient reported 0-10 analog pain scale, where 0 = no pain and 10 = worst pain imaginable. Reported as the change between timepoints.
Time Frame: Baseline (day 0), 45, 60, 75, 90, 105, 135, and 180 days
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Open Label Galcanezumab
Number analyzed (Participants) | 20
score on a scale
  Change from baseline to 60 days | -0.6224 (0.2663)
  Change from baseline to 90 days | -1.005 (0.2759)
  Change from baseline to 135 days | -0.8102 (0.2576)
  Change from baseline to 180 days | -1.079 (0.3816)
  Change from 45 days to 90 days | -0.3827 (0.2995)
  Change from 45 days to 135 days | -0.1877 (0.2796)
  Change from 45 days to 180 days | -0.4566 (0.3887)
  Change from 75 days to 135 days | 0.1949 (0.2876)
  Change from 75 days to 180 days | -0.07391 (0.3999)
  Change from 105 days to 180 days | -0.2689 (0.3922)

2. Primary Outcome: Number of Participants With a Change in Use of Anti-pain Medication
Description: Patient reported; any use of anti-pain medication.
Time Frame: Baseline through Day 135
Population: Data not collected on two participants who withdrew from the study. Two participants stopped one medication and started another.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Galcanezumab
Number analyzed (Participants) | 18
Participants
  Added one or more anti-pain medication | 3
  Stopped one or more anti-pain medication | 4
  No change | 13

3. Primary Outcome: Total Number of Adverse Events by Severity
Description: Recording all potential adverse events, based on lab results, patient side effects logs, patient vital sign measurement, and medical record review. Adverse events can be classified into five severity grades (1 = mild, 2 = moderate, 3 = severe, 4 = life threatening, and 5 = death).
Time Frame: Collected through Day 180
Measure: Number; unit: adverse events
Arm/Group | Open Label Galcanezumab
Number analyzed (Participants) | 20
adverse events
  1 = mild | 29
  2 = moderate | 5
  3 = severe | 0
  4 = life threatening | 0
  5 = death | 0

4. Secondary Outcome: Change in Level of TNF-alpha as a Marker of Pain or Inflammation
Description: Blood testing for presence of cytokine/chemokine pain or inflammation markers in patients' serum
Time Frame: Baseline, Day 180
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Open Label Galcanezumab
Number analyzed (Participants) | 20
pg/mL | 0.2 (0.3)

5. Secondary Outcome: Change in Level of IL-6 as a Marker of Pain or Inflammation
Description: Blood testing for presence of cytokine/chemokine pain or inflammation markers in patients' serum
Time Frame: Baseline, Day 180
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Open Label Galcanezumab
Number analyzed (Participants) | 20
pg/mL | 3.3 (4.2)

6. Other Pre Specified Outcome: Change in Circadian Rhythm Impairment
Description: Based on data from Wearable Sleep Monitor
Time Frame: Daily, from Baseline through Day 180
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Presence or Absence of DNA Polymorphisms That Predispose Treated Patients to Accentuated Responses of Either Lack of Response or Particularly Potent Response
Description: Genomic DNA testing
Time Frame: Day 0
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 180 days
Description: Patient adverse events were collected from week 4 week observation period to Day 180+/-3 days. Patients were systematically asked via patient diary and regular investigator assessments. Investigator assessments were administered at week 4 of observation period, day 30, day 45, phone call #1 between days 45 and 60, day 60, day 75, phone call #2 via days 75 and 90, day 105, day 135, and day 180. In addition, patient was able contact investigator or research coordinator in between assessments.
Arm/Group | Open Label Galcanezumab
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 13/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Galcanezumab (N=20)
Vomiting (Gastrointestinal disorders) | 1 — Unrelated
Urinary tract infection (Renal and urinary disorders) | 4 — Unrelated
Pain (Nervous system disorders) | 1 — Unrelated- had an attack of face pain and migraine headache
Dental caries (Infections and infestations) | 2 — Unrelated
Abdominal pain (Gastrointestinal disorders) | 1 — Unrelated
Numbness (Nervous system disorders) | 2 — Unrelated- one pt with tip of thumb tingling and another with tingling and numbness of hands(related to existing small fiber neuropathy)
Hypothyroidism (Endocrine disorders) | 1 — Unrelated
Insomnia (General disorders) | 1 — Related
Constipation (Gastrointestinal disorders) | 1 — Related
Vertigo (Ear and labyrinth disorders) | 1 — Unrelated
Fatigue (General disorders) | 1 — Unrelated
Fainting (Cardiac disorders) | 1 — Unrelated
Fall (General disorders) | 2 — Unrelated
Back pain (Injury, poisoning and procedural complications) | 1 — Unrelated-back injury causing back pain
Hypokalemia (General disorders) | 1 — Unrelated
Loss of awareness (Nervous system disorders) | 1 — Unrelated
Fracture (Injury, poisoning and procedural complications) | 1 — Unrelated
Dehydration (General disorders) | 1 — Unrelated
Elevated creatinine (Renal and urinary disorders) | 1 — Unrelated
Weight gain (General disorders) | 1 — Unrelated
Covid-19 infection (Infections and infestations) | 1 — Unrelated
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 — Related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT04158752/Prot_SAP_001.pdf